CLINICAL TRIAL: NCT00288769
Title: Oral Vitamin B12 as Potential Treatment of Recurrent Aphthous Stomatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: SOR415705CTIL
Record Dates: First submitted 2006-02-07; First posted 2006-02-08 (Estimated); Last update posted 2009-01-23 (Estimated); Status verified 2008-01

CONDITIONS: Recurrent Aphthous Stomatitis
Keywords: Recurrent aphthous stomatitis; vitamin B12
MeSH Terms: conditions — Stomatitis, Aphthous | interventions — Vitamin B 12

ARMS (1):
- 2 (Other)
  Interventions: Drug: daily sublingual tablets Vitamin B12 1000 mcg versus placebo

INTERVENTIONS:
Drug: daily sublingual tablets Vitamin B12 1000 mcg versus placebo

SUMMARY:
Background:

Recurrent aphthous stomatitis is a common phenomenon in Primary Medicine.Frequency of the phenomenon can be as high as 25% of the general population and the recurrence of the problem can be up to 50%.Different approaches for treatment are described: treatment with various natural vitamins , local ointments , disinfectant agents for local treatment , local antibiotic ointments , NSAID, local cortisone-steroids , and even medication on the basis of immune-depressants of the immune system and systematic steroids .

Methods:

A double-blind study of daily administration of sublingual Vitamin B12 tablets manufactured by Solgar (each tablet containing 1000 mcg. of Vitamin B12) opposed to placebo tablets.

Purpose of the research:

To investigate the effect of Vitamin B12 on the frequency of recurrent canker sores of the mouth (RAS).

Study hypothesis:

Treatment with vitamin B12 will reduce the recurrence rate and will diminish the symptomatology of RAS episodes.

DETAILED DESCRIPTION:
Scientific Background:

Recurrent painful canker sores within the mouth (Recurrent aphthous stomatitis, RAS) are a common phenomenon in Primary Medicine (1,2). The term "aphthai" in Greek means a condition within the mouth and is attributed to Hippocrates. (1) RAS is characterized by small, recurrent, painful canker sores in the mouth. These sores have characteristic round or elliptical ulcerations with sharp edges. The sores have a red halo surrounding them and a base with a yellowish or grey color (1,3). Frequency of the phenomenon can be as high as 25% of the general population and the recurrence of the problem can be up to 50% (2).

RAS is idiopathic in most cases. A possible cause is frequently a local injury or stress. Other possible causes include systemic illness, nutritional deficiency, sensitivity or allergy to certain foods, illness that effect the immune system and medication. Even though RAS can be associated with celiac disease or Behcet's disease, most of the cases patients are presented with this problem there is no other complaint or symptom and the patient is considered healthy.

Since the cause of the condition is unknown, Diagnosis is based on the patient's history and on a physical examination. There is no laboratory test that can substantiate or negate the condition (4-7).

In medical literature different approaches for treatment are described: treatment with various natural vitamins (8), local ointments (9), disinfectant agents for local treatment (10), local antibiotic ointments (11), non-steroidal anti-inflammatory ointments (NSAID)(12), local cortisone-steroids (13), and even medication on the basis of immune-depressants of the immune system and systematic steroids (14-16).

Most of these approaches that have been tried up to now have given temporary relief and only some have controlled the pain and healed the sores (16, 9-13).

In the past we have reported successfully treating three patients suffering from RAS with Vitamin B12 (17). We also have data regarding the treatment of 15 RAS patients. (This data has not yet been published.) The frequency of sores in this group had been an average of 1.5 episodes per month before treatment with Vitamin B12. During treatment the frequency decreased to 0.1 episode per month. As far as we know, there is no research using a double-blind design that investigated Vitamin B12 treatment of patients suffering from RAS.

Purpose of the research:

To investigate the effect of Vitamin B12 on the frequency of recurrent canker sores of the mouth (RAS).

Methods:

A double-blind study of daily administration of sublingual Vitamin B12 tablets manufactured by Solgar (each tablet containing 1000 mcg. of Vitamin B12, mannitol, stearic acid, Magnesium stearat , natural cherry flavor; weight of each tablet is 100 mcg.) opposed to placebo tablets (containing the same ingredients, except the Vitamin B12). The two types of tablets will be the same shape, size, color and have the same flavor. The tablets will be purchased from the Solgar Company in identical boxes, 30 tablets per box. The boxes will be numbered (1 or 2) - according to the type of treatment. The patient will receive instructions about daily treatment for a period of six (6) months, one tablet before going to sleep).

Sample Size:

In a retrospective study which we have done (to be published), we found that 73% of the patients who received Vitamin B12 there were no recurrent incidents of canker sores in the mouth. Assuming that among the patients that do not receive the Vitamin B12 treatment the frequency of the disease will be at least 90%, and that in the study group we expect that not more than 60% of the patients will continue to suffer from recurrent canker sores, in order to achieve a confidence level of 95% and a power of 80%, we need to recruit about 38 patients in the study group and 38 patients in the placebo group. With the assumption that the drop-out rate will be 30%, we need to recruit about 50 patients in each group.

Patients:

Candidates suffering from RAS who agree to participated in the study will sign a informed consent form.

Inclusion Criterion:

* Over 18 years old.
* Suffering from RAS as least for one year with a frequency of at least one sore per month.

Exclusion Criterion:

* Known systemic diseases concurrent with lesions in the mouth (Behcet's disease, Rheumatoid arthritis).
* Does not speak Hebrew, Russian, or English.
* Patients who have received in the last year Vit. B12 in any form.
* Patients who receive other treatment for RAS.
* Pregnant or nursing mothers.
* Patient known as suffering from Leber's optic atrophy.
* Patients suffering from psychosis.

Measurement for treatment effectiveness:

Principle measurement:

* Number of RAS occurrences during treatment (number of episodes per month).

Secondary measurements:

* Number of sores per RAS occurrence.
* Score of severity level according to a pain scale (Visual analog scale, VAS), average at time of RAS occurrence.

Measurement tools:

* Occurrence diary
* Pain Register

Research Design :

After receiving permission from the Helsinki Committee and before beginning the process of subject selection, we will register our research study with the International Clinical Registration System (/http://prsinfo.clinicaltrials.gov). Then we will recruit 20 primary physicians who will volunteer to ask 200 patients each concerning recurrent canker sores in the mouth. (These patients will be those who come to the physician for other reasons.) Out of these 4000 patients according to the literature, 800 patients suffer from RAS. We expect that half of these (about 400 patients) will report that the problem exists and half of those will agree to participate in the research study. According to our estimate, about 200 patients will adhere to the inclusion/exclusion criteria.

All the patients who are ready to participate in the study will receive from their physician the cell phone number of the Nose Throat and Ear physician (G.Z.) and the physician will ask the patient to contact G.Z. when they have a canker sore. In addition the patient's physician will also give the patient a written health synopsis, which will include any chronic diseases, sensitivity to medication and medical treatment. The patient will give this synopsis to one of the investigators ((IV, YP, RP, IR,) when they meet with him. The patient will then contact G.Z. and will be examined by him within 48 hours after the canker sore(s) appear to ascertain that the condition is actually recurrent aphthous stomatitis.

If the patient actually suffers from aphthous stomatitis, G.Z. will hand over the patient's information to one of the investigators. One of the investigators will contact the patient and make an appointment with him the next week.

Meetings with the patients:

One hundred (100) of the first patients who are found to suffer from aphthous stomatitis and who answer the inclusion/exclusion criteria will receive a detailed explanation in one of the languages, Hebrew, Russian, English about the purposes of the study, the research design, the risks involved in the research, and possible side effects. Those patients who sign the informed consent form will then be included in the study.

At this meeting the investigator will then fill out a form including socio-demographic data, a detailed anamnesis concerning the RAS (including number of years the patient has suffered from RAS, frequency of the problem in the past year, treatment that the patient has received for RAS in the past). The physician will also take measurements of height, weight and blood pressure.

The subjects will also have a blood test to measure the level of Vit. B12. (The sample will undergo centrifuge within the next few hours and the serum will be kept frozen until the test is done.) Since in our retrospective study (to be published) we did not find any difference in the result of treatment between people with patients having high and low levels of Vit. B12 in their blood, the level of Vit. B12 was not included as a criterion for inclusion or exclusion in the study.

The patients will receive instructions concerning filling out the "Canker Sore Diary" and the use of VAS. The patients will be given an appointment in another month. They will also receive the cell phone number for on of the investigators in order to contact him if and when an unexpected side effect occurs.

The subjects included in the study will be divided randomly into two groups (study group and control group).

Meetings with Research Assistant 1:

After a month from the time they met with the investigator, each patient will meet with Research Assistant 1 (physician), who will collect the "Canker Sore Diary" and will give the patient a bottle with 30 tablets of active ingredients or of placebo, according to which group he belongs (Control or Study). The patient will receive six (6) more appointments (once every month). The whole series of appointments will be decided in advance. A few days before each appointment the Research Assistant 1 will telephone the patient and remind him when and where the appointment will be.

During each of the six meetings the patient will give the Research Assistant 1 the "Canker Sore Diary", he will report on the new tablets that he has begun to take the last month, and the Research Assistant will count how many tablets are left in the bottle and will list the side effects, if any. At the end of the meeting the patient will receive the bottle of tablets for the next month.

In order to check the fact that the investigators did not know which patient was given which treatment, each investigator will be asked to "guess" which type of treatment each patient received.

Randomization:

Randomization was done by Research Assistant 2. Upon assigning a serial number for each subject, the Research Assistant will flip a coin according to which he will determine to which group the subject will belong. This number for the group will then be recorded on the form.

Assurance of "double blind" design: In order that the investigators will not know to which group the subject belongs, the code of the randomization will be saved in the computer in a protected by user name and the password will be know only to Research Assistant 2 (responsible for randomization, who will be the only one who knows in which box, No. 1 or No. 2, has the active ingredient, Vit. B12. The code which were assigned to the boxes for the investigators will be revealed only after the data has been processed. The research assistants will not take part in data processing.

Research Assistant 2 (responsible for randomization and knowing the code on the bottles) will not meet with the subjects and will not know any information about the subjects.

Statistical Analysis:

The data will be entered and processed by Research Assistant 3 in Epi-Info-Data 6.

Statistical Analysis will be done by the investigators with the aide of another research assistant (statistician) using SPSS. For statistical analysis the t-test and 2 will be used with a confidence level of P< 0.05.

References

1. Ship JA, Chavez EM, Doerr PA, Henson BS, Sarmadi M. Recurrent aphthous stomatitis. Quintessence Int 2000; 31:95-112.
2. Barrons RW. Treatment strategies for recurrent oral aphthous ulcers. Am J Health Syst Pharm 2001; 58:41-50.
3. Porter SR, Hegarty A, Kaliakatsou F, Hodgson TA, Scully C. Recurrent aphthous stomatitis. Clin Dermatol 2000; 18:569-78.
4. Piskin S, Sayan C, Durukan N, Senol M. Serum iron, ferritin, folic acid, and vitamin B12 levels in recurrent aphthous stomatitis. J Eur Acad Dermatol Venereol 2002; 16:66-7.
5. Wray D, Ferguson MM, Mason DK, Hutcheon AW, Dagg JH. Recurrent aphthae: treatment with vitamin B12, folic acid, and iron. BMJ 1975; 2:490-3.
6. Barnadas MA, Remacha A, Condomines J, de Moragas JM. [Hematologic deficiencies in patients with recurrent oral aphthae]. Med Clin (Barc) 1997; 109:85-7.
7. Natah SS, Konttinen YT, Enattah NS, Ashammakhi N, Sharkey KA, Hayrinen-Immonen R. Recurrent aphthous ulcers today: a review of the growing knowledge. Int J Oral Maxillofac Implants 2004; 33:221-34.
8. Pedersen A, Hougen HP, Klausen B, Winther K. LongoVital in the prevention of recurrent aphthous ulceration. J Oral Pathol Med 1990; 19:371-5.
9. Reznik D, O'Daniels CM. Clinical treatment evaluations of a new topical oral medication. Compend Contin Educ Dent Suppl 2001; 32:17-21.
10. Meiller TF, Kutcher MJ, Overholser CD, Niehaus C, DePaola LG, Siegel MA. Effect of an antimicrobial mouthrinse on recurrent aphthous ulcerations. Oral Surg Oral Med Oral Pathol Oral Radiol Endod 1991; 72:425-9.
11. Kerr AR, Drexel CA, Spielman AI. The efficacy and safety of 50 mg penicillin G potassium troches for recurrent aphthous ulcers. Oral Surg Oral Med Oral Pathol Oral Radiol Endod 2003; 96:685-94.
12. Murray B, McGuinness N, Biagioni P, Hyland P, Lamey PJ. A comparative study of the efficacy of Aphtheal in the management of recurrent minor aphthous ulceration. J Oral Pathol Med 2005; 34:413-9.
13. Gonzalez-Moles MA, Morales P, Rodriguez-Archilla A, Isabel IR, Gonzalez-Moles S. Treatment of severe chronic oral erosive lesions with clobetasol propionate in aqueous solution. Oral Surg Oral Med Oral Pathol Oral Radiol Endod 2002; 93:264-70.
14. Hutchinson VA, Angenend JL, Mok WL, Cummins JM, Richards AB. Chronic recurrent aphthous stomatitis: oral treatment with low-dose interferon alpha. Mol Biother 1990; 2:160-4.
15. Katz J, Langevitz P, Shemer J, Barak S, Livneh A. Prevention of recurrent aphthous stomatitis with colchicine: an open trial. J Am Acad Dermatol 1994; 31(3 Pt 1):459-61.
16. Femiano F, Gombos F, Scully C. Recurrent aphthous stomatitis unresponsive to topical corticosteroids: a study of the comparative therapeutic effects of systemic prednisone and systemic sulodexide. Int J Dermatol 2003; 42:394-7.
17. Volkov I, Rudoy I, Abu-Rabia U, Masalha T, Masalha R. Recurrent apthous stomatitis responsive to vitamin B12 treatment. Can Fam Phys 2005; 51:844-5.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old.
* Suffering from RAS as least for one year with a frequency of at least one sore per month

Exclusion Criteria:

* Known systemic diseases concurrent with lesions in the mouth (Behcet's disease, jaundice, Rheumatism, Aides).
* Does not speak Hebrew, Russian, or English.
* Patients who have received in the last year Vit. B12 in any form.
* Patients who receive other treatment for RAS.
* Pregnant or nursing mothers.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Dates: Start 2006-03; Primary Completion 2007-12 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ilia Volkov, MD, Principal Investigator — Ben-Gurion University of the Negev
Locations (1):
- Ben-Gurion University of the Negev, Beersheba, Israel

REFERENCES:
- [Result] Volkov I, Rudoy I, Freud T, Sardal G, Naimer S, Peleg R, Press Y. Effectiveness of vitamin B12 in treating recurrent aphthous stomatitis: a randomized, double-blind, placebo-controlled trial. J Am Board Fam Med. 2009 Jan-Feb;22(1):9-16. doi: 10.3122/jabfm.2009.01.080113. PMID 19124628